CLINICAL TRIAL: NCT00005000
Title: A Randomized, Open-Label, Study of Nelfinavir or Efavirenz in HIV-1 Infected, Antiretroviral Naive Patients
Brief Title: Treatment With Nelfinavir or Efavirenz of HIV-Infected Patients Who Have Never Received Anti-HIV Drugs
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Agouron Pharmaceuticals (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Model: Crossover | Purpose: Treatment
Other Study IDs: 259H; AG1343-1127
Record Dates: First submitted 2000-03-21; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-07

CONDITIONS: HIV Infections
Keywords: HIV-1; Drug Therapy, Combination; Lymphoid Tissue; HIV Protease Inhibitors; Genotype; Phenotype; Nelfinavir; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load; Adipose Tissue; Glucose; Lipids; Immunophenotyping; efavirenz
MeSH Terms: conditions — HIV Infections | interventions — Nelfinavir; efavirenz; Lamivudine; keyhole-limpet hemocyanin; Stavudine; Zidovudine; Didanosine

INTERVENTIONS:
Drug: Nelfinavir mesylate
Drug: Efavirenz
Drug: Lamivudine
Drug: Keyhole-Limpet Hemocyanin
Drug: Stavudine
Drug: Zidovudine
Drug: Didanosine

SUMMARY:
The purpose of this study is to compare two drugs (nelfinavir [NFV] and efavirenz [EFV]) used in start-up anti-HIV treatment. Doctors want to see if one is better than the other in extending the time that viral load (level of HIV in the blood) is kept low. The study will also look at the response of the immune system to each drug.

DETAILED DESCRIPTION:
Patients are randomized to initiate therapy and receive either nelfinavir (NFV) or efavirenz (EFV) in the first regimen (R1). All patients also receive zidovudine (AZT) and lamivudine (3TC). Patients are further randomized in a factorial fashion and by stratification based on HIV RNA level (less than 10,000, 10,000-100,000, or greater than 100,000 copies/ml) to be administered a single injection of a neo-antigen (KLH) at Week 12, 24, or 48. Therapy continues until switch criteria are met either before or after Week 24. When switch criteria are met, patients advance to the next regimen (R2).

R2 patients previously taking NFV switch to EFV; those randomized to EFV switch to NFV; the additional NRTIs change to stavudine (d4T) and didanosine (ddI). Therapy is continued for an additional 24 weeks.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this trial if they:

* Are HIV-positive.
* Have a CD4 count of at least 100 cells/mm3.
* Have a viral load of at least 5,000 copies/ml.

Exclusion Criteria

Patients may not be eligible for this study if they:

* Have taken any antiretroviral (anti-HIV) agent.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200
Dates: Start 1999-12

CONTACTS AND LOCATIONS:
Locations (1):
- Agouron Pharmaceuticals Inc, San Diego, California, United States